CLINICAL TRIAL: NCT00018096
Title: The Genetics of Environmental Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: John S. Sundy M.D., PhD., Duke University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NCRR-M01RR00030-0183; 2357
Record Dates: First submitted 2001-07-02; First posted 2001-07-04 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-05

CONDITIONS: Asthma
Keywords: Genetics; Lipopolysaccharide
MeSH Terms: conditions — Asthma | interventions — Sodium Chloride; Antigens, Dermatophagoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bronchoscopy (Experimental): 2 bronchoscopies 4 hours apart; The first to instill the 3 experimental biologic agents in separate airways (HDM, LPS and saline-placebo), the second to perform BAL and brush biopsies 4 hours later in the same airways.
  Interventions: Biological: LPS endotoxin, saline, HDM

INTERVENTIONS:
Biological: LPS endotoxin, saline, HDM — instillation of interventional products during bronchoscopy each down a different airway, each subject acts as their own control.
  Other Names: CCRE lipopolysaccharide endotoxin E.Coli O:113,Lot# 67801; House dust mite allergen (D.farinae) Greer Lab Lot #22574

SUMMARY:
In this project, we hypothesize that polymorphisms of genes expressed by the airway epithelia in asthmatics following specific airway challenges predispose individuals to the development of asthma. To test this hypothesis, we identify the genes that are differentially expressed by airway epithelial cells following challenge with stimuli that induce acquired (house dust mite) or innate (LPS) immune responses, and then determine whether polymorphisms in these genes are associated with the development of asthma in a separate, well characterized, familial cohort of asthmatics. This is a powerful approach that is designed to identify novel genes that are associated with both asthma pathogenesis (differentially expressed in the exposure-response study) and asthma susceptibility (genetically associated with asthma in a linkage/association study).

DETAILED DESCRIPTION:
The overall goal of this project is to identify genes that are involved in the development of airflow obstruction and airway inflammation in asthmatics, and to determine whether polymorphisms in these differentially expressed genes predispose individuals to develop asthma. Asthma is a complex genetic disorder that is caused by a number of unique gene-gene and gene-environment interactions. The search for asthma susceptibility genes has been complicated by the broad clinical phenotype of asthma, the polygenic inheritance pattern of this disease, and the substantial role of environmental exposures in the development and progression of asthma. Inhaled environmental agents induce several biologic responses in asthmatics; including the induction of acquired and innate immunity that leads to acute and chronic forms of airway inflammation and airway remodeling. Acquired immune responses to protein antigens, such as house dust mite allergen, often induce type 2 T lymphocyte-driven responses (Th2) which appear to be important in atopic asthma. Recent studies by our group and others demonstrate that innate immunity, initiated by inhalation of bacterial and viral pathogens, organic dusts, endotoxin or lipopolysaccharide (LPS), air pollution particulate matter, and ozone, can also cause acute and chronic forms of airflow obstruction, airway inflammation, and even airway remodeling. Emerging evidence indicates that both acquired and innate immune responses in the lung may be influenced by polymorphic genes. For instance, functional polymorphisms in the IL-4 receptor gene are thought to preferentially stimulate acquired Th2 immune responses to inhaled allergens, and we have recently shown that common co-segregating mutations in TLR4 (a transmembrane receptor for LPS) are associated with diminished airway responsiveness to inhaled LPS. These observations suggest that environmental challenges can be used to narrow the phenotype of asthma and investigate genetic susceptibility in biologically specific forms of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Atopic/asthmatic, atopic/non-asthmatic, non-atopic/asthmatic, or non-atopic/non-asthmatic
* Asthma subjects will be required to have either mild or moderate persistent asthma; positive methacholine challenge
* Atopic subjects should have seasonal allergy symptoms requiring medication and have positive skin test to house dust mite and at least 3 additional allergens. Serum IgE level >100.
* Willing/able to give informed consent & adhere to visit/protocol schedules.
* Screening visit laboratory, C-Xray, EKG, results within normal limits
* Women of childbearing potential must have a negative serum pregnancy test
* Screening Pulmonary Function testing above study criteria parameters

Exclusion Criteria:

* Systemic corticosteroid administration for asthma within the previous 90days
* Antibiotic administration within the previous 30 days.
* Viral respiratory infection within the previous 14 days.
* History of severe asthma requiring intubation.
* Occupational exposure to hay or grain dust.
* Significant exposure history to cigarette smoke
* Past or present history of allergen immunotherapy
* Underlying illnesses that may result in altered lung function
* Students or employees under direct supervision by protocol investigators are ineligible
* Subjects allergic to medications used (or potentially used) in the study will be excluded.
* Subjects using aspirin will be excluded
* Subjects who abuse alcohol or illicit substances will be excluded
* Medication use other than for asthma, allergies or contraception
* Other medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements
* Nursing mothers
* Other investigational medication within the last 30 days

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2001-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
BAL and endobronchial brush biopsy are measured and cell samples are analyzed to identify the genes in airway epithelia and inflammatory cells that are differentially expressed in response to LPS and dust mite antigen.RNA is isolated for gene expression. | 4 hours post first instillation bronchoscopy

SECONDARY OUTCOMES:
post bronchoscopy symptom followup | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sundy S. Sundy, MD. PhD., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States